CLINICAL TRIAL: NCT07273630
Title: Effect of Protein Supplementation and Fluid Restriction on Plasma Sodium Levels in Patients Undergoing Pituitary Surgery - a Randomized Open-label Active-controlled Trial -
Brief Title: Effect of Protein Supplementation and Fluid Restriction on Plasma Sodium Levels in Patients Undergoing Pituitary Surgery
Acronym: TREASURE-PIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-01549; kt25ChristCrain
Record Dates: First submitted 2025-11-14; First posted 2025-12-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Hyponatremia; Pituitary Surgery
Keywords: postoperative hyponatremia; hyponatremia; SIAD-related complications; protein supplementation; fluid restriction; Pituitary Surgery; Plasma Sodium Levels
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Limited fluid intake (Experimental): Patients will limit their total daily fluid intake
  Interventions: Dietary Supplement: Fluid restriction
- Additional protein (Experimental): Patients will consume additional protein daily
  Interventions: Dietary Supplement: Dietary protein supplementation
- No instructions (Active Comparator): Patients will not receive specific instructions.
  Interventions: Dietary Supplement: Standard post-operative care

INTERVENTIONS:
Dietary Supplement: Fluid restriction — Patients will limit their total daily fluid intake to a maximum of 1000 ml, including any liquids of their choice, such as water, milk, or juice.
  Arms: Limited fluid intake
Dietary Supplement: Dietary protein supplementation — Patients will consume an additional 80 grams of protein daily through two 150 ml protein drinks (40 grams of protein each, MOLTEIN PURE Drink, OMANDA) in various flavors. They can distribute the drinks throughout the day and drink other fluids freely based on thirst.
  Arms: Additional protein
Dietary Supplement: Standard post-operative care — Patients will not receive specific instructions on protein supplementation or fluid restriction. They will follow standard post-operative care and drink or eat freely based on natural appetite and thirst.
  Arms: No instructions

SUMMARY:
The investigators are conducting this study to investigate new preventive measures for patients with low sodium levels (hyponatremia), which can occur after surgery on the pituitary gland. This hyponatremia is often caused by the syndrome of inappropriate antidiuresis (SIAD). SIAD occurs when the pituitary gland secretes too much antidiuretic hormone. The antidiuretic hormone causes the kidneys to absorb more water. This dilutes the sodium in the blood and leads to hyponatremia. Low sodium levels are particularly common after pituitary surgery, as the procedure on the pituitary gland can lead to increased reactive secretion of antidiuretic hormone. At present, apart from educating patients about the symptoms of hyponatremia, there are no established standard measures for prevention after pituitary surgery. If hyponatremia is present, it is currently treated primarily by fluid restriction, which is not always pleasant or easy to adhere to. With this study, the investigators want to investigate whether protein supplementation or fluid restriction between day 4 and day 9 after surgery can serve as a preventive measure to stabilize sodium levels after pituitary surgery and improve the quality of life of patients.

DETAILED DESCRIPTION:
Disturbances in water balance, often due to disturbed arginine vasopressin (AVP) secretion from pituitary stalk and/or posterior lobe damage/manipulation, are common complications following pituitary surgery. This can result in either AVP deficiency, causing polyuria and polydipsia, or AVP excess, leading to water retention and dilutional hyponatremia (syndrome of inappropriate antidiuresis, SIAD). SIAD affects up to 30% of patients, typically developing between days 4 and 14 post-surgery, with a peak around day 7. While usually mild, severe hyponatremia is a leading cause of hospital readmission. Management includes fluid restriction, oral urea, or, in severe cases, hypertonic saline and AVP receptor antagonists.

Non-medicinal preventive strategies, such as prophylactic fluid restriction, have demonstrated efficacy in reducing SIAD incidence and hospital readmissions, but the optimal protocol remains unestablished. Dietary protein supplementation has recently emerged as a potential novel intervention, leveraging osmotic diuresis from increased endogenous urea production derived from the physiological amino-acid metabolism to raise plasma sodium levels. However, no data in the postoperative setting are available

This study aims to compare protein supplementation and fluid restriction to standard care (no specific intervention) in preventing post-pituitary surgery hyponatremia. From days 4 to 9 post-surgery, participants will receive one of the three treatments: Treatment A: Patients will limit their total daily fluid intake to a maximum of 1000 ml Treatment B: Patients will consume an additional 80 grams of protein daily through two 150 ml protein drinks (40 grams of protein each, MOLTEIN PURE Drink, OMANDA) in various flavors. Treatment C: Patients will not receive specific instructions. They will follow standard post-operative care and serve as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 or older) undergoing trans-sphenoidal or trans-cranial surgery for sellar / suprasellar pathology
* No pre-existing AVP-deficiency and SIAD or other causes of hyponatremia

Exclusion Criteria:

* AVP deficiency diagnosed before surgery based on established criteria
* Other type of neurosurgery / intracranial pathology / pre-existing spontaneous CSF -rhinorrhea
* Traumatic brain injury or intracranial hemorrhage
* Systemic infection or other causes for systemic stress
* Lactose intolerance, milk protein allergy, soy allergy, nuts allergy or known hypersensitivity or allergy to one of the components of the protein supplementation
* Inborn metabolic disorders implying carbohydrate, lipid, or protein metabolism
* Severe hepatic impairment (ALAT/ASAT >3x upper limit) or advanced symptomatic liver disease defined as past or current hepatic encephalopathy, liver cirrhosis Child C, or decompensated (bleeding, jaundice, hepatorenal syndrome)
* Reduction of eGFR <45 mL/min/1.73m² (KDIGO G3b, G4 and G5) or end stage renal disease (dialysis)
* Recently initiated (within the last 5 days) SGLT2 inhibitors, vaptans, or oral urea therapy
* Pregnancy or breastfeeding
* Lack of capacity or other reason preventing from giving informed consent or following study procedures.

Post-Inclusion Exclusion criteria (day 3 post-surgery, i.e.,time of randomization): - AVP deficiency diagnosed on post-operative day 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Odds ratio of treatment failure (intervention compared to standard of care) | 3 days post-surgery (time of randomization), and day 9 post-surgery.
  The primary objective is to evaluate the effectiveness of fluid restriction (Treatment A), and dietary protein supplementation (Treatment B) compared to the current standard care with no specific intervention and no fluid management guidance (Treatment C) in preventing treatment failure, defined at day 9 as a decrease in plasma sodium by at least 4 mmol/lL from baseline, and hyponatremia (plasma sodium <135mmol/L) or a decrease of at least 1 point in the MoCa score compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med., Principal Investigator — University Hospital Basel, Endocrinology
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided